CLINICAL TRIAL: NCT00637299
Title: Osteopathic Treatment May Improve Exercise Capacity in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Osteopathy in Chronic Obstructive Pulmonary Disease (COPD) Rehabilitation Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Ercole Zanotti, MD, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01/2008
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Results first posted 2009-04-20 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active osteopathic treatment (OMT+PR) (Active Comparator): The examination was performed by osteopathic practitioners with emphasis on the neuromusculoskeletal system including palpatory diagnosis for somatic dysfunction and viscerosomatic change, in the context of total patient care. The examination was concerned with range of motion of all parts of the body, performed with the patient in multiple positions to provide static and dynamic evaluation.
  Interventions: Other: Active osteopathic treatment (OMT+PR): Active Comparator
- SOT + PR (Sham Comparator): Sham osteopathic treatment (manipulation)
  Interventions: Other: sham osteopathic treatment (SOT+PR)

INTERVENTIONS:
Other: Active osteopathic treatment (OMT+PR): Active Comparator — The treatment was done once a week for 4 weeks and lasted 30 minutes.The examination was done according to the following scheme: anamnesis; physical examination (evaluation of the posture, palpation, tests for passive and active motion of areas linked to altered respiratory function); cranic-sacral evaluation (by means of a palpation of the cranic-sacral mechanism).
  Other Names: OMT+PR
  Arms: Active osteopathic treatment (OMT+PR)
Other: sham osteopathic treatment (SOT+PR) — Only soft manipulation was performed
  Other Names: SOT+PR
  Arms: SOT + PR

SUMMARY:
The purpose of this trial is to verify if an osteopathic treatment added to usual pulmonary rehabilitation trial is able to improve the walking ability of COPD patients and if there is any influence on lung functionality.

DETAILED DESCRIPTION:
The investigators decided to perform an osteopathic manipulative treatment (OMT) in a population of COPD patients. OMT was defined as the therapeutic application of manually guided forces by an osteopathic practitioner to improve physiologic function and/or support homeostasis that has been altered by somatic dysfunction. Concerning the respiratory system, osteopathy considers a model that describes the interdependent functions among five body components as follows: 1: the inherent motility of the brain and spinal cord; 2: fluctuation of the cerebrospinal fluid; 3: mobility of the intracranial and intraspinal membranes; 4: articular mobility of the cranial bones; 5: the involuntary mobility of the sacrum between the ilia. This model is the so called primary respiratory mechanism.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by COPD

Exclusion Criteria:

* other diseases other than COPD

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ercole Zanotti, md, Principal Investigator — Fondazione Salvatore Maugeri
Locations (1):
- Fondazione Salvatore Maugeri, Montescano, Pavia, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Osteopathic Treatment: OMT was defined as the therapeutic application of manually guided forces by an osteopathic practitioner.
- Sham Osteopathic Treatment (Manipulation): Sham Osteopathic Treatment was performed applying only soft manipulation
Period: Overall Study
Arm/Group | Active Osteopathic Treatment | Sham Osteopathic Treatment (Manipulation)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Osteopathic Treatment | Sham Osteopathic Treatment (Manipulation) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 12
  >=65 years | 2 | 6 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 64.2 (5.5) | 63.5 (4.7) | 63.8 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  Italy | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Walking Ability
Description: 6 minutes walking test (6MWT)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Active Osteopathic Treatment | Sham Osteopathic Treatment (Manipulation)
Number analyzed (Participants) | 10 | 10
meters | 369.5 (80) | 304.7 (96.6)
Statistical Analysis 1: Comparison: Active Osteopathic Treatment vs Sham Osteopathic Treatment (Manipulation); Test type: Superiority or Other; p < 0.01, t-test, 1 sided

2. Secondary Outcome: Lung Function Test
Description: residual volume (RV)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Active Osteopathic Treatment | Sham Osteopathic Treatment (Manipulation)
Number analyzed (Participants) | 10 | 10
liters | 3.09 (1.7) | 4.23 (1.4)
Statistical Analysis 1: Comparison: Active Osteopathic Treatment vs Sham Osteopathic Treatment (Manipulation); Test type: Superiority or Other; p < 0.05, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | Active Osteopathic Treatment | Sham Osteopathic Treatment (Manipulation)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No